CLINICAL TRIAL: NCT03247127
Title: The Memory Preservation Study of Whole Brain Radiotherapy With Hippocampal Avoidance for Patients With Brain Metastases
Brief Title: Memory Preservation of Hippocampal Avoidance Whole Brain Radiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KMUHIRB-E(II)20170081
Record Dates: First submitted 2017-07-27; First posted 2017-08-11 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Brain Metastases; Neurocognitive Function
Keywords: hippocampal avoidance whole brain radiotherapy (HA-WBRT); brain metastases; memory preservation; neurocognitive function
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Hippocampal avoidance -whole brain radiotherapy(HA-WBRT), which delivers radiation to whole brain and moreover, to reduce mean dose to hippocampal neural stem-cell compartment to minimize the neurocognitive function impairment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HA-WBRT (Other): Patients with brain metastases outside a 5-mm margin around either hippocampus and are eligible to this study will receive hippocampal avoidance whole brain radiotherapy 30 gray (Gy) in 10 fractions. The primary endpoint is Wechsler Memory Scale (Chinese) and cognitive abilities screening instrument (CASI) at 4 months.
  Interventions: Radiation: Hippocampal avoidance whole brain radiotherapy

INTERVENTIONS:
Radiation: Hippocampal avoidance whole brain radiotherapy — Planning target volume(PTV) for whole brain is Whole brain parenchyma plus2mm margin excluding metastases and HA region, 30Gy in 10 fractions will be delivered to PTVwhole brain. Bilateral Hippocampus will be contoured according to Radiation Therapy Oncology Group 0933 and hippocampal avoidance region is Hippocampi + 5mm margin. According to Radiation Therapy Oncology Group 0933 trial, dose to 100% of the hippocampus could not exceed 9 Gy, and maximal hippocampal dose could not exceed 16 Gy; dose to 100% of the hippocampus exceeding 10 Gy

SUMMARY:
The study aimed to investigate the memory preservation and neurocognitive function protection of hippocampal avoidance whole brain radiotherapy (HA-WBRT) among people who speak Mandarin Chinese or Taiwanese.

DETAILED DESCRIPTION:
Brain metastasis is very common, about 30% incidence rate for all patients with a diagnosis of cancer. The rising incidence of brain metastasis is most likely due to recent advances in systemic therapy, and use of magnetic resonance imaging (MRI). The most common primary site is the lung followed by breast. One of the standard treatments is whole brain radiotherapy; it can prolong the decline of neurocognitive function and improve quality of life. However, it can also cause decline in neurocognitive function as a late sequela. Memory impairment is the main cognitive function that affected by radiotherapy, and the neuronal stem cells located at hippocampal subgranular zone are highly sensitive to radiotherapy. There have been large randomized trials confirming that by HA-WBRT, the neurocognitive function decline can be reclaimed. In Taiwan, HA-WBRT is a popular and emerging treatment. However, not much study focused on its effects on neurocognitive function. The study is aimed to objectively investigate the memory preservation and neurocognitive function protection of HA-WBRT in people speaking Mandarin Chinese or Taiwanese by utilizing neurocognitive function test and QoL questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients with brain metastases, the brain metastases are located 5mm outside the hippocampus
* Pathologically proven diagnosis of nonhematopoietic malignancy other than germ cell malignancy
* No psychologic disorders
* Radiation Therapy Oncology Group recursive partitioning analysis class I or II
* First or second language: Mandarin Chinese or Taiwanese
* Signed the inform consensus

Exclusion Criteria:

* Less than 20 years old
* Leptomeningeal metastases or hydrocephalus
* Previous radiotherapy to head and neck region
* Creatinine >1.5mg/dl
* More than 2 extracranial metastases
* Patients who cannot tolerate memory or neurocognitive function test or cannot complete QoL questionnaire

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-03-27 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of Memory immediate recall and delayed recall | From baseline to 4 months after RT complete, tests are performed at baseline before radiotherapy begins, 2 months after radiotherapy complete and 4 months after radiotherapy complete.
  The memory battery is using Wechsler Memory Scale (Chinese), including Logical Memory I & II, Word Lists Ⅰ & II, Faces Ⅰ and spatial span.
Changes of general cognitive function | From baseline to 4 months after RT complete, tests are performed at baseline before radiotherapy begins, 2 months after radiotherapy complete and 4 months after radiotherapy complete.
  General cognitive function are tested using cognitive abilities screening instrument, CASI for screening and to test cognitive function as a whole.

SECONDARY OUTCOMES:
Changes of Quality of life | From baseline to 4 months after RT complete, the participants are requested to fill in the questionnaire of quality of life at baseline before radiotherapy begins, and 2 months after radiotherapy complete and 4 months after radiotherapy complete.
  Quality of life are assessed using The Functional Assessment of Cancer Therapy-Brain (FACT-Br) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Pen-Tzu Fang, MD, Principal Investigator — Department of Radiation Oncology, Kaohsiung Medical University Hospital
Locations (1):
- Fang, Pen-Tzu, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gondi V, Pugh SL, Tome WA, Caine C, Corn B, Kanner A, Rowley H, Kundapur V, DeNittis A, Greenspoon JN, Konski AA, Bauman GS, Shah S, Shi W, Wendland M, Kachnic L, Mehta MP. Preservation of memory with conformal avoidance of the hippocampal neural stem-cell compartment during whole-brain radiotherapy for brain metastases (RTOG 0933): a phase II multi-institutional trial. J Clin Oncol. 2014 Dec 1;32(34):3810-6. doi: 10.1200/JCO.2014.57.2909. Epub 2014 Oct 27. PMID 25349290
- [Result] Aoyama H, Tago M, Kato N, Toyoda T, Kenjyo M, Hirota S, Shioura H, Inomata T, Kunieda E, Hayakawa K, Nakagawa K, Kobashi G, Shirato H. Neurocognitive function of patients with brain metastasis who received either whole brain radiotherapy plus stereotactic radiosurgery or radiosurgery alone. Int J Radiat Oncol Biol Phys. 2007 Aug 1;68(5):1388-95. doi: 10.1016/j.ijrobp.2007.03.048. PMID 17674975
- [Result] Roman DD, Sperduto PW. Neuropsychological effects of cranial radiation: current knowledge and future directions. Int J Radiat Oncol Biol Phys. 1995 Feb 15;31(4):983-98. doi: 10.1016/0360-3016(94)00550-8. PMID 7860415
- [Result] DeAngelis LM, Delattre JY, Posner JB. Radiation-induced dementia in patients cured of brain metastases. Neurology. 1989 Jun;39(6):789-96. doi: 10.1212/wnl.39.6.789. PMID 2725874
- [Result] Ghia A, Tome WA, Thomas S, Cannon G, Khuntia D, Kuo JS, Mehta MP. Distribution of brain metastases in relation to the hippocampus: implications for neurocognitive functional preservation. Int J Radiat Oncol Biol Phys. 2007 Jul 15;68(4):971-7. doi: 10.1016/j.ijrobp.2007.02.016. Epub 2007 Apr 18. PMID 17446005
- [Result] Gondi V, Tome WA, Marsh J, Struck A, Ghia A, Turian JV, Bentzen SM, Kuo JS, Khuntia D, Mehta MP. Estimated risk of perihippocampal disease progression after hippocampal avoidance during whole-brain radiotherapy: safety profile for RTOG 0933. Radiother Oncol. 2010 Jun;95(3):327-31. doi: 10.1016/j.radonc.2010.02.030. Epub 2010 Apr 12. PMID 20392503
- [Result] Gondi V, Tolakanahalli R, Mehta MP, Tewatia D, Rowley H, Kuo JS, Khuntia D, Tome WA. Hippocampal-sparing whole-brain radiotherapy: a "how-to" technique using helical tomotherapy and linear accelerator-based intensity-modulated radiotherapy. Int J Radiat Oncol Biol Phys. 2010 Nov 15;78(4):1244-52. doi: 10.1016/j.ijrobp.2010.01.039. PMID 20598457
- [Result] Gutierrez AN, Westerly DC, Tome WA, Jaradat HA, Mackie TR, Bentzen SM, Khuntia D, Mehta MP. Whole brain radiotherapy with hippocampal avoidance and simultaneously integrated brain metastases boost: a planning study. Int J Radiat Oncol Biol Phys. 2007 Oct 1;69(2):589-97. doi: 10.1016/j.ijrobp.2007.05.038. PMID 17869672